CLINICAL TRIAL: NCT04352608
Title: A Randomized, Double-Blinded, Placebo-Controlled, Phase Ⅰ/Ⅱ Clinical Trial, to Evaluate the Safety and Immunogenicity of the SARS-CoV-2 Inactivated Vaccine in Healthy Adults Aged 18~59 Years
Brief Title: Safety and Immunogenicity Study of Inactivated Vaccine for Prophylaxis of SARS CoV-2 Infection (COVID-19)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sinovac Research and Development Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Sinovac Biotech Co., Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PRO-nCOV-1001
Record Dates: First submitted 2020-04-14; First posted 2020-04-20 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2021-07

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (12):
- Emergency schedule & Two doses of medium dosage vaccine (Experimental): 24 participants in phase Ⅰand 60 participants in phase Ⅱ will receive two doses of medium dosage inactivated SARS-CoV-2 vaccine at the emergency vaccination schedule,and 60 participants in phase Ⅱ will receive one dose of booster immunization with medium dosage vaccine 6 months after the emergency schedule
  Interventions: Biological: Two doses of medium dosage inactivated SARS-CoV-2 vaccine at the emergency vaccination schedule
- Emergency schedule & Two doses of high dosage vaccine (Experimental): 24 participants in phase Ⅰand 60 participants in phase Ⅱ will receive two doses of high dosage inactivated SARS-CoV-2 vaccine at the emergency vaccination schedule,and 60 participants in phase Ⅱ will receive one dose of booster immunization with high dosage vaccine 6 months after the emergency schedule
  Interventions: Biological: Two doses of high dosage inactivated SARS-CoV-2 vaccine at the emergency vaccination schedule
- Emergency schedule &Two doses of placebo (Placebo Comparator): 24 participants in phase Ⅰand 30 participants in phase Ⅱ will receive two doses of placebo at the emergency vaccination schedule,and 30 participants in phase Ⅱ will receive one dose of booster immunization with placebo 6 months after the emergency schedule
  Interventions: Biological: Two doses of placebo at the emergency vaccination schedule
- Routine schedule & Two doses of medium dosage vaccine (Experimental): 24 participants in phase Ⅰand 60 participants in phase Ⅱ will receive two doses of medium dosage inactivated SARS-CoV-2 vaccine at the routine vaccination schedule,and 60 participants in phase Ⅱ will receive one dose of booster immunization with medium dosage vaccine 6 months after the routine schedule
  Interventions: Biological: Two doses of medium dosage inactivated SARS-CoV-2 vaccine at the routine vaccination schedule
- Routine schedule &Two doses of high dosage vaccine (Experimental): 24 participants in phase Ⅰand 60 participants in phase Ⅱ will receive two doses of high dosage inactivated SARS-CoV-2 vaccine at the routine vaccination schedule,and 60 participants in phase Ⅱ will receive one dose of booster immunization with high dosage vaccine 6 months after the routine schedule
  Interventions: Biological: Two doses of high dosage inactivated SARS-CoV-2 vaccine at the routine vaccination schedule
- Routine schedule & Two doses of placebo (Placebo Comparator): 24 participants in phase Ⅰand 30 participants in phase Ⅱ will receive two doses of placebo at the routine vaccination schedule,and 30 participants in phase Ⅱ will receive one dose of booster immunization with placebo 6 months after the routine schedule
  Interventions: Biological: Two doses of placebo at the routine vaccination schedule
- Emergency schedule & Three doses of medium dosage vaccine (Experimental): 60 participants in phase Ⅱ will receive three doses of medium dosage inactivated SARS-CoV-2 vaccine at the emergency vaccination schedule
  Interventions: Biological: Three doses of medium dosage inactivated SARS-CoV-2 vaccine at the emergency vaccination schedule
- Emergency schedule & Three doses of high dosage vaccine (Experimental): 60 participants in phase Ⅱ will receive three doses of high dosage inactivated SARS-CoV-2 vaccine at the emergency vaccination schedule
  Interventions: Biological: Three doses of high dosage inactivated SARS-CoV-2 vaccine at the emergency vaccination schedule
- Emergency schedule &Three doses of placebo (Placebo Comparator): 30 participants in phase Ⅱ will receive three doses of placebo at the emergency vaccination schedule
  Interventions: Biological: Three doses of placebo at the emergency vaccination schedule
- Routine schedule & Three doses of medium dosage vaccine (Experimental): 60 participants in phase Ⅱ will receive three doses of medium dosage inactivated SARS-CoV-2 vaccine at the routine vaccination schedule
  Interventions: Biological: Three doses of medium dosage inactivated SARS-CoV-2 vaccine at the routine vaccination schedule
- Routine schedule &Three doses of high dosage vaccine (Experimental): 60 participants in phase Ⅱ will receive three doses of high dosage inactivated SARS-CoV-2 vaccine at the routine vaccination schedule
  Interventions: Biological: Three doses of high dosage inactivated SARS-CoV-2 vaccine at the routine vaccination schedule
- Routine schedule &Three doses of placebo (Placebo Comparator): 30 participants in phase Ⅱ will receive three doses of placebo at the routine vaccination schedule
  Interventions: Biological: Three doses of placebo at the routine vaccination schedule

INTERVENTIONS:
Biological: Two doses of medium dosage inactivated SARS-CoV-2 vaccine at the emergency vaccination schedule — Two doses of medium dosage (600SU/0.5ml) experimental vaccine at the schedule of day 0,14,and one dose of booster immunization with medium dosage (600SU/0.5ml) experimental vaccine 6 months after the schedule of day 0,14 in phaseⅡ.
  Arms: Emergency schedule & Two doses of medium dosage vaccine
Biological: Two doses of high dosage inactivated SARS-CoV-2 vaccine at the emergency vaccination schedule — Two doses of high dosage (1200 SU/0.5ml) experimental vaccine at the schedule of day 0,14 and one dose of booster immunization with high dosage (1200SU/0.5ml) experimental vaccine 6 months after the schedule of day 0,14 in phaseⅡ.
  Arms: Emergency schedule & Two doses of high dosage vaccine
Biological: Two doses of placebo at the emergency vaccination schedule — Two doses of placebo at the schedule of day 0,14 and one dose of booster immunization with placebo 6 months after the schedule of day 0,14 in phaseⅡ.
  Arms: Emergency schedule &Two doses of placebo
Biological: Two doses of medium dosage inactivated SARS-CoV-2 vaccine at the routine vaccination schedule — Two doses of medium dosage (600SU/0.5ml) experimental vaccine at the schedule of day 0,28 and one dose of booster immunization with medium dosage (600SU/0.5ml) experimental vaccine 6 months after the schedule of day 0,28 in phaseⅡ.
  Arms: Routine schedule & Two doses of medium dosage vaccine
Biological: Two doses of high dosage inactivated SARS-CoV-2 vaccine at the routine vaccination schedule — Two doses of high dosage (1200 SU/0.5ml) experimental vaccine at the schedule of day 0,28 and one dose of booster immunization with high dosage (1200SU/0.5ml) experimental vaccine 6 months after the schedule of day 0,28 in phaseⅡ
  Arms: Routine schedule &Two doses of high dosage vaccine
Biological: Two doses of placebo at the routine vaccination schedule — Two doses of placebo at the schedule of day 0,28 and one dose of booster immunization with placebo 6 months after the schedule of day 0,28 in phaseⅡ.
  Arms: Routine schedule & Two doses of placebo
Biological: Three doses of medium dosage inactivated SARS-CoV-2 vaccine at the emergency vaccination schedule — Three doses of medium dosage (600SU/0.5ml) experimental vaccine at the schedule of day 0,14,42
  Arms: Emergency schedule & Three doses of medium dosage vaccine
Biological: Three doses of high dosage inactivated SARS-CoV-2 vaccine at the emergency vaccination schedule — Three doses of high dosage (1200 SU/0.5ml) experimental vaccine at the schedule of day 0,14,42
  Arms: Emergency schedule & Three doses of high dosage vaccine
Biological: Three doses of placebo at the emergency vaccination schedule — Three doses of placebo at the schedule of day 0,14,42
  Arms: Emergency schedule &Three doses of placebo
Biological: Three doses of medium dosage inactivated SARS-CoV-2 vaccine at the routine vaccination schedule — Three doses of medium dosage (600SU/0.5ml) experimental vaccine at the schedule of day 0,28,56
  Arms: Routine schedule & Three doses of medium dosage vaccine
Biological: Three doses of high dosage inactivated SARS-CoV-2 vaccine at the routine vaccination schedule — Three doses of high dosage (1200 SU/0.5ml) experimental vaccine at the schedule of day 0,28,56
  Arms: Routine schedule &Three doses of high dosage vaccine
Biological: Three doses of placebo at the routine vaccination schedule — Three doses of placebo at the schedule of day 0,28,56
  Arms: Routine schedule &Three doses of placebo

SUMMARY:
This study is a randomized, double-blinded, and placebo controlled phase Ⅰ/Ⅱ clinical trial of the SARS-CoV-2 inactivated vaccine manufactured by Sinovac Research & Development Co., Ltd. The purpose of this study is to evaluate the safety and immunogenicity of the experimental vaccine in healthy adults aged 18~59 Years.

DETAILED DESCRIPTION:
This study is a randomized, double-blinded, single-center, placebo-controlled phase Ⅰ/Ⅱ clinical trial in adults aged 18~59 years. The purpose of this study is to evaluate the immunogenicity and safety of the experimental SARS-CoV-2 inactivated vaccine. The experimental vaccine and placebo were both manufactured by Sinovac Research & Development Co., Ltd. A total of 744 subjects will be enrolled, with 144 at phase Ⅰ, and 600 at phase Ⅱ. All of participants in phase Ⅰ will be assigned to receive two doses of experimental vaccine or placebo on the schedule of day 0,14 or day 0,28.300 participants in phase Ⅱ will be assigned to receive two doses of experimental vaccine or placebo on the schedule of day 0,14 or day 0,28 and one dose of booster immunization will be given 6 months after primary immunization of day 0,14 or day 0,28.The other 300 participants in phase Ⅱ will be assigned to receive three doses of experimental vaccine or placebo on the schedule of day 0,14,42 or 0,28,56 .

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18-59 years;
* Proven legal identity;
* Participants should be capable of understanding the informed consent form, and such form should be signed prior to enrolment ;

Exclusion Criteria:

* Travel history / residence history of Wuhan city and surrounding areas, or other communities with case reports within 14 days;
* History of contact with a SARS-CoV-2 infection (positive in nucleic acid test) within 14 days;
* Have contacted patients with fever or respiratory symptoms from Wuhan and surrounding areas, or from communities with case reports within 14 days;
* Have contacted patients with fever or respiratory symptoms from Wuhan and surrounding areas, or from communities with case reports within 14 days;
* Self-reported history of SARS;
* Self-reported history of new coronavirus infection;
* Positive in serum antibodies (IgG or IgM) screening of COVID-19;
* Positive in nasopharyngeal swabs or anal swabs through RT-PCR;
* Women who are breastfeeding, pregnant or planning to become pregnant during the study period;
* BMI≥35 kg/m2;
* History of asthma, history of allergy to the vaccine or vaccine components, or serious adverse reactions to the vaccine, such as urticaria, dyspnea, and angioedema;
* Congenital malformations or developmental disorders, genetic defects, severe malnutrition, etc.;
* Autoimmune disease or immunodeficiency / immunosuppression;
* Suffering from severe chronic diseases, severe cardiovascular diseases, hypertension and diabetes that cannot be controlled by drugs, liver and kidney diseases, malignant tumors, etc.;
* Severe neurological disease (epilepsy, convulsions or convulsions) or mental illness;
* Thyroid disease or history of thyroidectomy, spleenlessness, functional spleenlessness, spleenlessness or splenectomy resulting from any condition;
* Diagnosed abnormal blood coagulation function (eg, lack of blood coagulation factors, blood coagulopathy, abnormal platelets) or obvious bruising or blood coagulation;
* Immunosuppressive therapy, cytotoxic therapy, inhaled corticosteroids (excluding allergic rhinitis corticosteroid spray therapy, acute non-complicated dermatitis superficial corticosteroid therapy) in the past 6 months;
* Abnormal laboratory test results in the physical examination such as clinically significant abnormal hematology and biochemistry beyond the reference value range (only applicable to Phase I clinical trials);
* History of alcohol or drug abuse;
* Receipt of blood products within in the past 3 months;
* Receipt of other investigational drugs in the past 30 days;
* Receipt of attenuated live vaccines in the past 14 days;
* Receipt of inactivated or subunit vaccines in the past 7 days;
* Attacks of acute diseases or chronic diseases in the past 7 days;
* Axillary temperature >37.0°C;
* According to the investigator's judgment, the subject has any other factors that are not suitable for participating in the clinical trial.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 744 (Actual)
Dates: Start 2020-04-16 (Actual); Primary Completion 2020-07-10 (Actual); Study Completion 2021-07-24 (Actual)

PRIMARY OUTCOMES:
Safety indexes of adverse reactions | From Day 0 to Day 28 after each dose
  Incidence of adverse reactions occured from Day 0 to Day 28 after each dose
Immunogenicity indexes of neutralizing-antibody seroconversion rates | The 14th day /the 28th day after two doses of vaccination
  The seroconversion rate of neutralizing antibodies 14 days (emergency schedule)/28 days (routine schedule) after the two-dose vaccination.

SECONDARY OUTCOMES:
Safety indexes of adverse reactions | 7 days after each dose of vaccination
  Incidence of adverse reactions 7 days after each dose of vaccination
Safety indexes of Incidence of abnormal laboratory index | On the 3th day after each dose of vaccination in phase Ⅰ
  Incidence of abnormal laboratory index (blood routine test, blood chemistry test,and urine routine test) on the 3th day after each dose of vaccination in phase Ⅰ
Safety indexes of serious adverse events (SAEs） | From the beginning of the vaccination to 6 months post the whole-schedule vaccination
  Incidence of SAEs from the beginning of the vaccination to 6 months post the whole-schedule vaccination
Immunogenicity indexes of the seropositive rate, GMT, and GMI of neutralizing antibodies | 14 days (emergency schedule)/28 days (routine schedule) after two-dose vaccination
  The seropositive rate, GMT, and GMI of neutralizing antibodies 14 days (emergency schedule)/28 days (routine schedule) after two-dose vaccination
Immunogenicity indexes of the seroconversion rate, seropositive rate, GMT and GMI of neutralizing antibodies | 28 days after the two doses (emergency schedule)
  The seroconversion rate, seropositive rate, GMT and GMI of neutralizing antibodies 28 days after the two doses (emergency schedule)
Immunogenicity indexes of the seroconversion rate, seropositive rate, GMT, and GMI in Phase Ⅱ | 28 days after the third dose （only for days 0,14,42 and days 0,28,56 schedule）
  Phase Ⅱ:The seroconversion rate, seropositive rate, GMT, and GMI 28 days after the third dose（only for days 0,14,42 and days 0,28,56 schedule）
Immunogenicity indexes of the seropositivity rate, GMT, and GMI in Phase Ⅱ | 14 day (emergency schedule)/28 days (routine schedule) after the booster dose （only for days 0,14 and days 0,28 schedule）
  Phase Ⅱ:The seropositivity rate, GMT, and GMI 14 day (emergency schedule)/28 days (routine schedule) after the booster dose （only for days 0,14 and days 0,28 schedule）
Immunogenicity indexes of the seroconversion rate, seropositive rate, GMT, and GMI in Phase Ⅰ | 7/14/21 days after the first dose vaccination (emergency schedule)
  Phase Ⅰ:The seroconversion rate, seropositive rate, GMT, and GMI 7/14/21 days after the first dose vaccination (emergency schedule)
Immunogenicity indexes of the seroconversion rate, seropositive rate, GMT, and GMI in Phase Ⅰ | 28/35/42 days after the first dose vaccination (routine schedules)
  Phase Ⅰ:The seroconversion rate, seropositive rate, GMT, and GMI 28/35/42 days after the first dose vaccination (routine schedules)
Immunogenicity indexes of the seropositive rate of IgG, IgM antibodies | 7/14/21/28/42 days after the first dose vaccination (emergency schedule)
  Phase Ⅰ:The seropositive rate of IgG, IgM antibodies 7/14/21/28/42 days after the first dose vaccination (emergency schedule)
Immunogenicity indexes of the seropositive rate of IgG,IgM antibodies | 28/35/42/56 days after the first dose vaccination (routine schedule)
  Phase Ⅰ: The seropositive rate of IgG,IgM antibodies 28/35/42/56 days after the first dose vaccination (routine schedule)

CONTACTS AND LOCATIONS:
Overall Officials: Fengcai Zhu, Doctor, Principal Investigator — Jiangsu Provincial Center for Disease Control and Prevention
Locations (1):
- Suining County Center for Disease Control and Prevention, Xuzhou, Jiangsu, China

REFERENCES:
- [Derived] Xin Q, Wu Q, Chen X, Han B, Chu K, Song Y, Jin H, Chen P, Lu W, Yang T, Li M, Zhao Y, Pan H, Yu H, Wang L. Six-month follow-up of a booster dose of CoronaVac in two single-centre phase 2 clinical trials. Nat Commun. 2022 Jun 3;13(1):3100. doi: 10.1038/s41467-022-30864-w. PMID 35660738
- [Derived] Zeng G, Wu Q, Pan H, Li M, Yang J, Wang L, Wu Z, Jiang D, Deng X, Chu K, Zheng W, Wang L, Lu W, Han B, Zhao Y, Zhu F, Yu H, Yin W. Immunogenicity and safety of a third dose of CoronaVac, and immune persistence of a two-dose schedule, in healthy adults: interim results from two single-centre, double-blind, randomised, placebo-controlled phase 2 clinical trials. Lancet Infect Dis. 2022 Apr;22(4):483-495. doi: 10.1016/S1473-3099(21)00681-2. Epub 2021 Dec 8. PMID 34890537
- [Derived] Zhang Y, Zeng G, Pan H, Li C, Hu Y, Chu K, Han W, Chen Z, Tang R, Yin W, Chen X, Hu Y, Liu X, Jiang C, Li J, Yang M, Song Y, Wang X, Gao Q, Zhu F. Safety, tolerability, and immunogenicity of an inactivated SARS-CoV-2 vaccine in healthy adults aged 18-59 years: a randomised, double-blind, placebo-controlled, phase 1/2 clinical trial. Lancet Infect Dis. 2021 Feb;21(2):181-192. doi: 10.1016/S1473-3099(20)30843-4. Epub 2020 Nov 17. PMID 33217362